CLINICAL TRIAL: NCT03883633
Title: Reversal of Cognitive Decline (ReCODE) Study
Acronym: RECODE
Status: Completed | Type: Observational
Sponsor: QuesGen Systems Inc (Other)
Responsible Party: Sponsor
Other Study IDs: RECODE-1018
Record Dates: First submitted 2019-03-13; First posted 2019-03-21 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-03

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Dementia; Alzheimer's Disease; Cognitive Decline; MCI
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrolled Participants: All participants enrolled will be tracked from initial assessment to study completion.
  Interventions: Behavioral: ReCODE Protocol

INTERVENTIONS:
Behavioral: ReCODE Protocol — Functional medicine approach to address symptoms of Alzheimer's and cognitive decline
  Other Names: Bredesen Protocol

SUMMARY:
Prospective study on patients enrolled in the ReCODE treatment protocol

DETAILED DESCRIPTION:
The objective of the study is to determine if the ReCODE treatment has a measurable impact on the typical progression of neurocognitive decline observed in patients with Alzheimer's Disease (AD) and patients who are exhibiting Mild Cognitive Impairment (MCI). MCI is often a precursor to an AD diagnosis. For this study, there will be no distinction made between participants who have been diagnosed with AD and those who show signs of MCI.

ELIGIBILITY:
Inclusion Criteria:

* 45 to 76 years old
* Adults of any gender, race or ethnicity
* Subjects must have cognitive impairment as demonstrated by a combination of AQ-21 over 5 and either a MOCA 26 or below or a CNS Vitals screening assessment in the MCI in the bottom 70th percentile or 2 of the subtests in the bottom 50th percentile.
* Proficient in spoken and written English for consenting as well as for study participation.
* Must be able to use a computer and web interface. If assistance is needed, it must be readily available to them.
* Regular access to a computer and an internet connection since certain aspects of the program (e.g. cognitive training) are delivered electronically
* Willing and able to follow the protocol if the treating physician determines that is required for appropriate patient care.

Exclusion Criteria:

* Uncontrolled major medical illness, seizures, cardiovascular or cerebrovascular instability.
* A major psychiatric diagnosis that affects activities of daily living (ADL) or functioning.
* Currently taking psychoactive medications known to impact cognition.
* Use of statin therapy, unless eligible to discontinue.
* Use of anticoagulation therapy or history of deep vein thrombosis.
* MRI findings of hydrocephalus, focal stroke, extensive white matter disease or brain tumor.
* Experienced Traumatic Brain Injury (TBI) that is severe enough that it has an ongoing impact on patient function on a regular basis.
* Lack of support (either family member or caregiver) to assist with following the treatment protocol.
* Active cancer, cancer within the past five years or any history of breast cancer.
* Inability to exercise.
* Inability to use a computer, or no computer access.
* Unwillingness or ineligibility to use bioidentical hormone replacement.
* Pregnancy or any chance of becoming pregnant during the course of the study period.
* Presence of an existing diagnosis of a non-AD neurodegenerative disorder (e.g., Lewy Body Disease, Frontotemporal Disease, Chronic Traumatic Encephalopathy, Korsakoff's Syndrome).
* Diagnosis of cerebrovascular disease as the primary cause of cognitive impairment.
* Previous treatment or experience with ReCODE.

Ages: 45 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who have signs of reduced neurocognitive function
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in short-time memory function | Given at enrollment and repeated at three months, six months and nine months after enrollment
  Participants will be given an on-line assessment to test memory and recall using CNS (Central Nervous System) Vitals assessment.
Changes in cognitive function | Given at enrollment and repeated at three months, six months and nine months after enrollment
  Participants will be evaluated for cognitive capability using the Montreal Cognitive Assessment (MoCA)
Perceived changes in capability assessed by input from care giver or family member | Given at enrollment and repeated at three months, six months and nine months after enrollment
  Care givers will be surveyed about the participants capability using an assessment based on the Alzheimer's Questionnaire 21-question assessment (AQ-21)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Hathaway, MD, Principal Investigator — Ann Hathaway MD; Deborah Gordon, MD, Principal Investigator — Northwest Memory Center; Kat Toups, MD, Principal Investigator — Kat Toups MD
Locations (3):
- United States (3):
  - Ann Hathaway MD, San Rafael, California
  - Bay Area Wellness, Walnut Creek, California
  - Northwest Memory Center, Ashland, Oregon

IPD SHARING:
Plan to Share IPD: No